CLINICAL TRIAL: NCT00296400
Title: Randomised, Double-blind, 52-wk, Parallel-grp Multicentre, PIIb Study to Evaluate Effects of Rosuvastatin 10mg, Rosuvastatin 40mg and Atorvastatin 80mg on Urinary Protein Excretion in Hypercholesterolaemic Non-diabetic Patients With Moderate Proteinuria
Brief Title: Prospective Evaluation of Proteinuria and Renal Function in Non-diabetic Patients With Progressive Renal Disease
Acronym: PLANET II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3569C00011; PLANET II
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Results first posted 2010-12-30 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; Proteinuria; Diabetes Mellitus
MeSH Terms: conditions — Hyperlipidemias; Proteinuria; Diabetes Mellitus | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
Drug: Atorvastatin

SUMMARY:
The purpose of this study is to evaluate the effects of Crestor (rosuvastatin) and (Lipitor) atorvastatin on urinary protein excretion over 1 year in non-diabetes with moderate proteinuria and hypercholesterolaemia.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* Hyperlipidemia
* Urinary protein

Exclusion Criteria:

* Previous rosuvastatin treatment < 6 months prior to Visit 1
* Statin intolerance
* Severe hypertension
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Crestor Medical Science Director, MD, Study Director — AstraZeneca
Locations (107):
- United States (23):
  - Research Site, Avondale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Pasadena, California
  - Research Site, Riverside, California
  - Research Site, Clearwater, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Topeka, Kansas
  - Research Site, Columbia, Maryland
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Columbia, Missouri
  - Research Site, Orchard Park, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Gig Harbor, Washington
  - Research Site, Milwaukee, Wisconsin
- Brazil (2):
  - Research Site, Curitiba, Paraná
  - Research Site, São Paulo, São Paulo
- Bulgaria (8):
  - Research Site, Blagoevgrad
  - Research Site, Burgas
  - Research Site, Gabrovo
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Canada (12):
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Courtice, Ontario
  - Research Site, East York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Richmond Hill, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Denmark (6):
  - Research Site, Copenhagen
  - Research Site, Fredericia
  - Research Site, Herlev
  - Research Site, Holbæk
  - Research Site, Roskilde
  - Research Site, Viborg
- Germany (8):
  - Research Site, Berlin
  - Research Site, Cloppenburg
  - Research Site, Demmin
  - Research Site, Düsseldorf
  - Research Site, Elsenfeld
  - Research Site, Göttingen
  - Research Site, Hanover
  - Research Site, Würzburg
- Hungary (14):
  - Research Site, Ajka
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Gy�r
  - Research Site, Keszthely
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szolnok
  - Research Site, Szombathely
  - Research Site, Zalaegerszeg
- Italy (14):
  - Research Site, Bergamo, BG
  - Research Site, Bologna, BO
  - Research Site, Brescia, BS
  - Research Site, Acireale, CT
  - Research Site, Foggia, FG
  - Research Site, Florence, FI
  - Research Site, Parma, PR
  - Research Site, Reggio Calabria, RC
  - Research Site, Sassari, SS
  - Research Site, Teramo, TE
  - Research Site, Torino, TO
  - Research Site, Castelfranco Veneto, TV
  - Research Site, Treviso, TV
  - Research Site, Mestre, VE
- Mexico (7):
  - Research Site, Zapopan, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, D.F, Mexico
  - Research Site, San Luis Potos�, Mexico
  - Research Site, Cuernavaca, Morelos
  - Research Site, Aguascalientes
  - Research Site, Durango
- Romania (8):
  - Research Site, Brasov, Brașov County
  - Research Site, Cluj-Napoca, Cluj
  - Research Site, Constanța, Constanța County
  - Research Site, Suceava, Suceava
  - Research Site, Timișoara, Timiș County
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Iași
- South Africa (5):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Pretoria, South Africa
  - Research Site, Parow, W Cape
  - Research Site, Cape Town
  - Research Site, Durban

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] de Zeeuw D, Anzalone DA, Cain VA, Cressman MD, Heerspink HJ, Molitoris BA, Monyak JT, Parving HH, Remuzzi G, Sowers JR, Vidt DG. Renal effects of atorvastatin and rosuvastatin in patients with diabetes who have progressive renal disease (PLANET I): a randomised clinical trial. Lancet Diabetes Endocrinol. 2015 Mar;3(3):181-90. doi: 10.1016/S2213-8587(14)70246-3. Epub 2015 Feb 4. PMID 25660356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 797 patients entered the study with moderate proteinuria and hypercholesterolemia and were receiving stable treatment with angiotensin converting enzyme (ACE) inhibitors and/or angiotensin receptor blockers (ARBs) for 3 or more months prior to Visit 1. The study was conducted at 114 participating centers in 11 countries.
Pre-assignment Details: 237 patients [pts] completed the 8-week lead-in period and were randomized. The most common reasons for discontinuation during the lead in period included incorrect enrollment (466 pts), development of study-specific discontinuation criteria (41 pts), and voluntary discontinuation (29 pts). 189 patients completed the study.
Period: Overall Study
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Started | 70 | 87 | 80
Completed | 53 | 69 | 67
Not Completed | 17 | 18 | 13
Not completed — Adverse Event | 7 | 7 | 7
Not completed — Withdrawal by Subject | 5 | 6 | 2
Not completed — Incorrect enrollment | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Study specific discontinuation criteria | 0 | 0 | 1
Not completed — Visit 10 was performed earlier | 0 | 1 | 0
Not completed — Pregnancy | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg | Total
Number analyzed (Participants) | 70 | 87 | 80 | 237
Age, Customized [Number; unit: Participants]
  18 to 49 years | 34 | 44 | 42 | 120
  50 to 64 years | 31 | 31 | 30 | 92
  >=65 years | 5 | 12 | 8 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 [lower limit 28] | 35 [lower limit 35] | 31 [lower limit 31] | 94 [0 to 0]
  Male | 42 [lower limit 42] | 52 [lower limit 52] | 49 [lower limit 49] | 143 [0 to 0]
Estimated glomerular filtration rate [eGFR] [Mean (Standard Deviation); unit: mL/min] | 78.315 (28.0653) [78.315 to 28.03653] | 76.774 (30.3878) [76.774 to 30.3878] | 71.464 (30.0156) [71.464 to 30.0156] | 75.419 (29.6012) [0 to 88.43993]
Urine albumin/creatinine ratio [Mean (Standard Deviation); unit: mg/g] | 1023.165 (720.0251) [1023.165 to 720.0251] | 1167.368 (865.4584) [1167.368 to 865.4584] | 1069.103 (720.8011) [1069.103 to 720.8011] | 1091.263 (775.1889) [0 to 2306.2846]
Urine protein/creatinine ratio [Mean (Standard Deviation); unit: mg/g] | 1301.163 (832.7398) [1301.163 to 832.7398] | 1487.131 (1068.0642) [1487.131 to 1068.0642] | 1439.720 (991.2295) [1439.720 to 991.2295] | 1416.023 (975.7636) [0 to 2892.0335]

OUTCOME MEASURES:

1. Primary Outcome: Urinary Protein/Creatinine Ratio at Week 52 [LOCF]
Description: Urinary protein/creatinine ratio (mg/g) =urine protein concentration (mg/dL)/ urine creatinine concentration (g/dL). Outcome measure is the ratio of Week 52 [LOCF] urine protein/creatinine ratio over baseline urine protein/creatinine ratio.
Time Frame: Assessed at baseline and Week 52 (LOCF)
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 65 | 80 | 75
ratio | 0.938 [0.725 to 1.212] | 1.082 [0.927 to 1.262] | 0.759 [0.636 to 0.905]

2. Secondary Outcome: Urinary Protein/Creatinine Ratio at Week 26.
Description: Urinary protein/creatinine ratio (mg/g) =urine protein concentration (mg/dL)/ urine creatinine concentration (g/dL). Outcome measure is the ratio of Week 26 urine protein/creatinine ratio over baseline urine protein/creatinine ratio.
Time Frame: Assessed at baseline and Week 26
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 59 | 76 | 70
ratio | 0.932 [0.721 to 1.203] | 1.057 [0.898 to 1.244] | 0.762 [0.631 to 0.921]

3. Secondary Outcome: Urinary Albumin/Creatinine Ratio at Week 26
Description: Urinary albumin/creatinine ratio (mg/g) =urine albumin concentration (mg/dL)/ urine creatinine concentration (g/dL). Outcome measure is the ratio of Week 26 urine albumin/creatinine ratio over baseline urine albumin/creatinine ratio.
Time Frame: Assessed at baseline and Week 26
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 60 | 76 | 72
ratio | 0.850 [0.631 to 1.143] | 0.946 [0.789 to 1.135] | 0.731 [0.601 to 0.889]

4. Secondary Outcome: Urinary Albumin/Creatinine Ratio at Week 52 [LOCF]
Description: Urinary albumin/creatinine ratio (mg/g) =urine albumin concentration (mg/dL)/ urine creatinine concentration (g/dL). Outcome measure is the ratio of Week 52 [LOCF] urine albumin/creatinine ratio over baseline urine albumin/creatinine ratio.
Time Frame: Assessed at baseline and Week 52 [LOCF]
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 65 | 80 | 75
ratio | 0.879 [0.652 to 1.185] | 0.967 [0.814 to 1.148] | 0.719 [0.587 to 0.882]

5. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 26
Description: The change from baseline in eGFR at Week 26 is the Week 26 value minus baseline value.
Time Frame: Assessed at baseline and Week 26
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 60 | 77 | 72
mL/min | 1.39 (15.431) [lower limit 15.431] | -3.41 (13.228) [lower limit 13.228] | -1.61 (9.494) [lower limit 9.494]

6. Secondary Outcome: Change From Baseline in eGFR at Week 52 [LOCF]
Description: The change from baseline in eGFR at Week 52 [LOCF] is the Week 52 value or last observation carried forward minus baseline value.
Time Frame: Assessed at baseline and Week 52 [LOCF]
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 65 | 80 | 75
mL/min | -2.71 (13.083) [lower limit 13.083] | -3.30 (12.325) [lower limit 12.325] | -1.74 (13.964) [lower limit 13.964]

7. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in Total Cholesterol [TC] at Week 26.
Description: Correlation of changes from baseline in urinary protein/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 26. (Correlation values range from -1 to +1. -1 indicates a perfect negative linear relationship while a +1 indicates a perfect linear positive relationship. A value of zero indicates no relationship.)
Time Frame: baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Groups:
- Rosuvastatin: Rosuvastatin Treatments pooled
- Atorvastatin: Atorvastatin Treatment
- All Treatments: All Treatments pooled
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 135 | 70 | 205
Correlation coefficient | 0.17601 | 0.21701 | 0.19643

8. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in Total Cholesterol [TC] at Week 52.
Description: Correlation of changes from baseline in urinary protein/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 52. (Correlation values range from -1 to +1. -1 indicates a perfect negative linear relationship while a +1 indicates a perfect linear positive relationship. A value of zero indicates no relationship.)
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 64 | 185
Correlation coefficient | 0.20462 | 0.03480 | 0.16077

9. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 26
Description: as for outcome 7
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 135 | 69 | 204
Correlation coefficient | 0.14302 | 0.24393 | 0.17632

10. Secondary Outcome: Correlation of Changes From Baseline inUrinary Protein/Creatinine Ratio With Percent Change From Baseline in LDL-C
Description: as for outcome 8
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 62 | 183
Correlation coefficient | 0.16868 | -0.09428 | 0.10679

11. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in High Density Lipoprotein Cholesterol [HDL-C] at Week 26
Description: as for outcome 7
Time Frame: 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 135 | 69 | 204
Correlation coefficient | 0.18055 | 0.24987 | 0.22094

12. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in HDL-C at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 62 | 183
Correlation coefficient | 0.20346 | 0.18041 | 0.20818

13. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in Non-high Density Lipoprotein Cholesterol [nonHDL-C] at Week 26
Description: Correlation of changes from baseline in urinary protein/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 26. (Correlation values range from -1 to +1. -1 indicates a perfect negative linear relationship while a +1 indicates a perfect linear positive relationship. A value of zero indicates no relationship.
  )
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 135 | 69 | 204
Correlation coefficient | 0.16206 | 0.20032 | 0.17628

14. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in nonHDL-C at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 62 | 183
Correlation coefficient | 0.20386 | -0.04698 | 0.14495

15. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in Triglyceride [TG] at Week 26
Description: as for outcome 7
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 135 | 70 | 205
Correlation coefficient | 0.15348 | -0.06049 | 0.10089

16. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in TG at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 64 | 185
Correlation coefficient | 0.20659 | 0.23989 | 0.21728

17. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in TC/HDL-C Ratio at Week 26
Description: as for outcome 7
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 135 | 69 | 204
Correlation coefficient | 0.04652 | 0.06344 | 0.04149

18. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in TC/HDL-C Ratio at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 62 | 183
Correlation coefficient | 0.03957 | -0.17644 | -0.01549

19. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in LDL-C/HDL-C Ratio at Week 26
Description: as for outcome 7
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 135 | 69 | 204
Correlation coefficient | 0.06383 | 0.12687 | 0.07462

20. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in LDL-C/HDL-C Ratio at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 62 | 183
Correlation coefficient | 0.05881 | -0.20262 | -0.01340

21. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in nonHDL-C/HDL-C Ratio at Week 26
Description: as for outcome 7
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 135 | 69 | 204
Correlation coefficient | 0.06794 | 0.05410 | 0.05465

22. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in nonHDL-C/HDL-C Ratio at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 62 | 183
Correlation coefficient | 0.07188 | -0.16669 | 0.00955

23. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in Apolipoprotein A-1 [ApoA-1] at Week 26
Description: as for outcome 7
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 131 | 67 | 198
Correlation coefficient | 0.12595 | 0.05628 | 0.13754

24. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in ApoA-1 at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 62 | 178
Correlation coefficient | 0.19626 | 0.09835 | 0.18349

25. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in Apolipoprotein B [ApoB] at Week 26
Description: as for outcome 7
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 131 | 67 | 198
Correlation coefficient | 0.18504 | 0.17259 | 0.19146

26. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in ApoB at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 62 | 178
Correlation coefficient | 0.18473 | -0.02690 | 0.12496

27. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in ApoB/ApoA-1 Ratio at Week 26
Description: as for outcome 7
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 131 | 67 | 198
Correlation coefficient | 0.10698 | 0.13814 | 0.11414

28. Secondary Outcome: Correlation of Changes From Baseline in Urinary Protein/Creatinine Ratio With Percent Change From Baseline in ApoB/ApoA-1 Ratio at Week 52
Description: as for outcome 8
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 62 | 178
Correlation coefficient | 0.05859 | -0.12938 | -0.00540

29. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in TC at Week 26
Description: Correlation of changes from baseline in urinary albumin/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 26. (Correlation values range from -1 to +1. -1 indicates a perfect negative linear relationship while a +1 indicates a perfect linear positive relationship. A value of zero indicates no relationship.)
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 136 | 72 | 208
Correlation coefficient | 0.18188 | 0.17503 | 0.18566

30. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in TC at Week 52
Description: Correlation of changes from baseline in urinary albumin/creatinine ratio with percent change from baseline in lipids and lipoprotein concentrations at Week 52. (Correlation values range from -1 to +1. -1 indicates a perfect negative linear relationship while a +1 indicates a perfect linear positive relationship. A value of zero indicates no relationship.)
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 65 | 186
Correlation coefficient | 0.23734 | 0.01311 | 0.17958

31. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in LDL-C at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 136 | 71 | 207
Correlation coefficient | 0.14783 | 0.21561 | 0.16899

32. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in LDL-C at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | 0.20285 | -0.13565 | 0.12568

33. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in HDL-C at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 136 | 71 | 207
Correlation coefficient | 0.23547 | 0.25043 | 0.25208

34. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in HDL-C at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | 0.17479 | 0.18677 | 0.18203

35. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in nonHDL-C at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 136 | 71 | 207
Correlation coefficient | 0.16080 | 0.17150 | 0.16578

36. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in nonHDL-C at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | 0.24107 | -0.08640 | 0.16525

37. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in TG at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 136 | 72 | 208
Correlation coefficient | 0.11526 | -0.06890 | 0.07248

38. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in TG at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 65 | 186
Correlation coefficient | 0.21730 | 0.21151 | 0.21477

39. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in TC/HDL-C Ratio at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 136 | 71 | 207
Correlation coefficient | 0.02506 | 0.02201 | 0.01860

40. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in TC/HDL-C Ratio at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | 0.08954 | -0.20870 | 0.01926

41. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in LDL-C/HDL-C Ratio at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 136 | 71 | 207
Correlation coefficient | 0.05037 | 0.09779 | 0.05936

42. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in LDL-C/HDL-C Ratio at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | 0.10365 | -0.24717 | 0.01386

43. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in nonHDL-C/HDL-C Ratio at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 136 | 71 | 207
Correlation coefficient | 0.04955 | 0.02740 | 0.03798

44. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in nonHDL-C/HDL-C Ratio at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | 0.11997 | -0.21073 | 0.03955

45. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in ApoA-1 at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 131 | 68 | 199
Correlation coefficient | 0.16499 | 0.02609 | 0.15049

46. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in ApoA-1 at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 63 | 179
Correlation coefficient | 0.20021 | 0.12953 | 0.18870

47. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in ApoB at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 131 | 68 | 199
Correlation coefficient | 0.18720 | 0.16167 | 0.18717

48. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in ApoB at Week 52
Description: as for outcome 30
Time Frame: 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 63 | 179
Correlation coefficient | 0.21082 | -0.04379 | 0.14085

49. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in ApoB/ApoA-1 Ratio at Week 26
Description: as for outcome 29
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 131 | 68 | 199
Correlation coefficient | 0.10258 | 0.13505 | 0.11103

50. Secondary Outcome: Correlation of Changes From Baseline in Urinary Albumin/Creatinine Ratio With Percent Change From Baseline in ApoB/ApoA-1 Ratio at Week 52
Description: as for outcome 30
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 63 | 179
Correlation coefficient | 0.08108 | -0.16753 | 0.00479

51. Secondary Outcome: Correlation of Changes From Baseline in eGFR With Percent Change From Baseline in TC at Week 26
Description: Correlation of changes from baseline in eGFR with percent change from baseline in lipids and lipoprotein concentrations at Week 26. (Correlation values range from -1 to +1. -1 indicates a perfect negative linear relationship while a +1 indicates a perfect linear positive relationship. A value of zero indicates no relationship.)
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 137 | 72 | 209
Correlation coefficient | 0.06641 | -0.07964 | 0.02900

52. Secondary Outcome: Correlation of Changes From Baseline in eGFR With Percent Change From Baseline in TC at Week 52
Description: Correlation of changes from baseline in eGFR with percent change from baseline in lipids and lipoprotein concentrations at Week 52. (Correlation values range from -1 to +1. -1 indicates a perfect negative linear relationship while a +1 indicates a perfect linear positive relationship. A value of zero indicates no relationship.)
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 65 | 186
Correlation coefficient | -0.15721 | 0.16110 | -0.05794

53. Secondary Outcome: Correlation of Changes From Baseline in eGFR With Percent Change From Baseline in LDL-C at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 137 | 71 | 208
Correlation coefficient | 0.02679 | -0.07603 | -0.00171

54. Secondary Outcome: Correlation of Changes From Baseline in eGFR With Percent Change From Baseline in LDL-C at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | -0.15731 | 0.15368 | -0.06310

55. Secondary Outcome: Correlation of Changes From Baseline in eGFR With Percent Change From Baseline in HDL-C at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 137 | 71 | 208
Correlation coefficient | 0.01684 | 0.01755 | 0.01758

56. Secondary Outcome: Correlation of Changes From Baseline in eGFR With Percent Change From Baseline in HDL-C at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | 0.14080 | 0.02750 | 0.09472

57. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in nonHDL-C at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 137 | 71 | 208
Correlation coefficient | 0.06029 | -0.08151 | 0.02283

58. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in nonHDL-C at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | -0.19532 | 0.14967 | -0.09001

59. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in TG at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 137 | 72 | 209
Correlation coefficient | 0.04160 | 0.00531 | 0.03430

60. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in TG
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 65 | 186
Correlation coefficient | -0.12643 | 0.00486 | -0.08301

61. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in TC/HDL-C Ratio at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 137 | 71 | 208
Correlation coefficient | 0.08194 | -0.06576 | 0.04477

62. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in TC/HDL-C Ratio at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | -0.23597 | 0.19933 | -0.10205

63. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in LDL-C/HDL-C Ratio at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 137 | 71 | 208
Correlation coefficient | 0.04858 | -0.05535 | 0.02023

64. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in LDL-C/HDL-C Ratio at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | -0.20805 | 0.18299 | -0.07681

65. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in nonHDL-C/HDL-C Ratio at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 137 | 71 | 208
Correlation coefficient | 0.08263 | -0.06860 | 0.04337

66. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in nonHDL-C/HDL-C Ratio at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 121 | 63 | 184
Correlation coefficient | -0.23887 | 0.17170 | -0.10817

67. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in ApoA1 at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 132 | 68 | 200
Correlation coefficient | 0.13029 | 0.17554 | 0.14191

68. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in ApoA1 at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 63 | 179
Correlation coefficient | 0.11047 | 0.07751 | 0.08580

69. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in ApoB at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 132 | 68 | 200
Correlation coefficient | 0.06098 | -0.03181 | 0.03861

70. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in ApoB at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 63 | 179
Correlation coefficient | -0.11217 | 0.11006 | -0.03932

71. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in ApoB/ApoA-1 Ratio at Week 26
Description: as for outcome 51
Time Frame: Baseline and 26 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 132 | 68 | 200
Correlation coefficient | 0.02907 | -0.09476 | -0.00160

72. Secondary Outcome: Correlation of Change From Baseline in eGFR With Percent Change From Baseline in ApoB/ApoA-1 Ratio at Week 52
Description: as for outcome 52
Time Frame: Baseline and 52 weeks
Measure: Number; unit: Correlation coefficient
Arm/Group | Rosuvastatin | Atorvastatin | All Treatments
Number analyzed (Participants) | 116 | 63 | 179
Correlation coefficient | -0.15415 | 0.10486 | -0.06121

ADVERSE EVENTS:
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Serious Adverse Events (participants affected / at risk) | 10/69 | 6/87 | 5/80
Other Adverse Events (participants affected / at risk) | 15/69 | 16/87 | 17/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10 mg (N=69) | Rosuvastatin 40 mg (N=87) | Atorvastatin 80 mg (N=80)
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypertensive Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Intracranial Aneurysm (Nervous system disorders) | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10 mg (N=69) | Rosuvastatin 40 mg (N=87) | Atorvastatin 80 mg (N=80)
Nausea (Gastrointestinal disorders) | 2 | 6 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 7
Bronchitis (Infections and infestations) | 4 | 0 | 0
Blood Creatine Phosphokinase Increased (Infections and infestations) | 3 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5
Dizziness (Nervous system disorders) | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less